CLINICAL TRIAL: NCT04808427
Title: Magnetic Resonance Image (MRI) Guided High Energy Ultrasound for Focal Prostate Cancer Ablation
Brief Title: Pilot Study to Investigate Magnetic Resonance (MR) Image Guided Focal Therapy in Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210017; 21-C-0017
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11-24

CONDITIONS: Prostate Cancer
Keywords: TULSA; Thermal Therapy System; PSA; Gleason Score
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 1/Arm 1 (Experimental): Ultrasound ablation of focal prostate cancer
  Interventions: Device: TULSA-PRO

INTERVENTIONS:
Device: TULSA-PRO — Transurethral MR-Thermometry Guided Ultrasound Ablation of the Prostate

SUMMARY:
Background:

The ability to treat early prostate cancer is still limited. Thermal ablation methods are being tested for focal prostate cancer therapy. Researchers want to improve on these methods.

Objective:

To understand if Transurethral UltraSound Ablation (TULSA) in combination with MRI guidance is useful to treat localized prostate cancer.

Eligibility:

English-speaking adults ages 18 and older with localized prostate cancer that can be seen on MRI and can be treated by thermal ablation.

Design:

Participants will be screened with the following:

* Medical history
* Physical exam
* Digital rectal exam
* Blood and urine tests
* Electrocardiogram
* Tumor biopsy
* Questionnaire to assess urinary tract symptoms
* MRI of the pelvis. The MRI scanner is a long, narrow tube. Participants will lie on a bed that moves in and out of the scanner.

Participants may also be screened with the following:

* Echocardiogram
* Chest x-ray
* Bone scan
* Urodynamic studies to see how well the bladder, sphincters, and urethra hold and release urine
* MRI of the brain
* Transrectal ultrasound
* Computer tomography (CT) scan of the chest, abdomen, and pelvis. A CT scan is a series of x-ray images taken of parts of the body.

Some screening tests will be repeated during the study.

Participants will have the TULSA procedure. They will have an MRI for guidance. A small ultrasound applicator will be placed into their urethra. It uses heat to destroy the cancer areas in the prostate. It is controlled by a robotic arm. A cooling catheter will be placed into their rectum.

Participants will use a urethral catheter for 1-7 days.

Participants will have follow-up visits at 3, 6, 12, 18, 24, and 36 months.

DETAILED DESCRIPTION:
Background:

Prostate cancer is relatively slow growing, with doubling times for local tumors estimated at 2 to 4 years.

Some prostate cancers prove to be small, low grade, and noninvasive and they appear to pose little risk to the life or health of the host. Recent patient series suggest that 20% to 30% of men undergoing radical prostatectomy have pathologic features in the radical prostatectomy specimen consistent with an insignificant or "indolent" cancer which poses little threat to life or health.

We propose that participants with low volume and low grade disease can be best served with focal ablation of the visible prostate cancer without the side effects of urinary incontinence and erectile dysfunction associated with radiation therapy or radical surgery.

Focal Therapy for prostate cancer has gained popularity however prior studies demonstrate a failure rate as high as 50% with a laser.

Objective:

To determine the feasibility of magnetic resonance image (MRI)-guided ultrasound-induced thermal therapy of biopsy-confirmed and MRI visible, prostate tumor(s) using the TULSA Thermal Therapy System (Profound Medical)

Eligibility:

Subjects with prostate cancer, amenable for ultrasound ablation

Organ confined clinical T1c or clinical T2a prostate cancer, visible on MRI, and confirmed by prostate biopsy

Adequate organ and marrow function

Prostate-specific antigen (PSA) < 20 ng/ml

Age >=18 years

Design:

Study testing feasibility and tolerability of ultrasound ablation of focal prostate cancer.

It is anticipated that 15 participants will be evaluated for this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must have prostate cancer amenable for ultrasound ablation defined as:

* diagnosed by transrectal ultrasound-guided prostate biopsy via standard 12 core biopsy and targeted biopsy of any MRI-visible or tracked lesions; pathological diagnosis must be confirmed by Laboratory of Pathology, NCI;
* Gleason Score <= 7;
* MRI-visible or MRI-tracked prostate cancer. This includes prostate cancer found on targeted biopsy of MRI-visible or MRI-tracked lesion. Histologically positive standard biopsy cores of Grade Group >= 2 prostate cancer must be from an area overlying or within 1cm of an MRI-visible or tracked lesion(s) and reviewed by NCI urologic pathologist. (Left / Right, Base, Mid-Gland, Apex). Systematic and targeted cores of Grade Group 1 prostate cancer outside of proposed ablation zone do not affect inclusion status, as these can be observed by conventional guideline management.
* organ confined clinical T1c or clinical T2a prostate cancer that is visualized on MRI. Note: Participants after prostate cancer treatment with local recurrence or residual tumor which is visible on MRI are eligible.
* PSA < 20 ng/ml or PSA >20 with a PSA density <0.15.
* Adults (>= 18 years of age)
* Participants must have adequate organ and marrow function as defined below:

Platelets >= 50,000/mcL

Hemoglobin >= 8 g/dL

Measured or calculated creatinine clearance (CrCl) (eGFR may also be used in place of CrCl)* >= 30 mL/min/1.73 m^2

GFR=glomerular filtration rate; ULN=upper limit of normal.

*Creatinine clearance (CrCl) or eGFR should be calculated per institutional standard.

* Subjects must be able to understand and willing to sign a written informed consent document.
* Subjects must be co-enrolled to NCI protocol 16-C-0010 "Care of the Prostate Cancer Patient and Prospective Procurement of Prostate Cancer Tissue."

EXCLUSION CRITERIA:

* Targeted lesion ablation length from apex to base of >5 cm or lesion extending >3 cm from the urethra.
* Target ablation volume greater than 100 ml.
* Presence of calcifications that would impede ultrasound transmission between the urethra and ablative target.
* Participants are unable to tolerate MRI (foreign body, i.e., pacemaker or other implanted device; claustrophobia; inability to tolerate rectal coil; etc.)
* Acute urinary tract infection
* Lower urinary tract symptoms defined by an IPSS > 20
* Participants with uncontrolled coagulopathies (including liver dysfunction, or untreated hereditary coagulopathies which have a standard of care treatment) per surgeon discretion based on bleeding risk.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation (within time frame) that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
feasibility and tolerability | 3, 6, 12, 18, 24, and 36 months
  To determine the feasibility of magnetic resonance image (MRI)-guided ultrasound-induced thermal therapy of biopsy-confirmed and MRI visible, prostate tumor(s) using the TULSA Thermal Therapy System (Profound Medical)

SECONDARY OUTCOMES:
safety and tolerability | 3, 6, 12, 18, 24, and 36 months
  Address short- and long-term complication rates of study treatment by tabulating adverse events by grade according to CTCAE, and analyzing and reporting descriptively
changes in imaging and biopsy characteristics | 3, 6, 12, 18, 24, and 36 months
  Determine if focal ablation of MRI visible, biopsy-confirmed prostate cancer using the TULSA Thermal Therapy System (Profound Medical) platform can successfully ablate targeted prostate cancer lesions in >50% of participants
effect of thermal ablation on short- and long-term complication rates | 3, 6, 12, 18, 24, and 36 months
  Observe thermal damage on post-contrast MRI which extends into areas of the Rectum or Urethra; assess frequency of not completing the procedure
thermal damage | 3, 6, 12, 18, 24, and 36 months
  Observe thermal damage on post-contrast MRI which extends into areas of the Rectum or Urethra; assess frequency of not completing the procedure
outcome of TULSA ablation | 3, 6, 12, 18, 24, and 36 months
  Use descriptive statistical analysis to examine serial PSA, PSA density, changes in imaging and biopsy, International Prostate Symptom Score (IPSS), and Sexual Health Inventory for Men (SHIM)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0017.html